CLINICAL TRIAL: NCT00417066
Title: The Flexible GnRH Antagonist Protocol Provides Better Results (IVF Outcomes) Than Flare up GnRH Agonist Protocol in Poor Responders
Brief Title: Flexible GnRH Antagonist vs Flare up GnRH Agonist Protocol in Poor Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eugonia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: poor responders
Record Dates: First submitted 2006-12-22; First posted 2006-12-29 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-01

CONDITIONS: Infertility; Premature Ovarian Failure
Keywords: poor responders; GnRH antagonist; GnRH agonist; flare up; short protocol
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency | interventions — ganirelix; Triptorelin Pamoate

INTERVENTIONS:
Drug: Ganirelix 0.25mg (Orgalutran, Organon, The Netherlands)
Drug: Arvekap 0.1mg (Triptorelin, Ipsen, France)

SUMMARY:
The purpose of this study is to compare ovulation induction using a flexible GnRH antagonist protocol and flare up GnRH agonist protocol in IVF patients with poor response to ovarian stimulation. Our hypothesis is that the antagonist protocol provides better IVF outcomes compared to the flare up protocol in this group of patients.

DETAILED DESCRIPTION:
Poor responders are women who fail to respond effectively to the usual gonadotropin stimulation protocol applied in an IVF cycle. It seems that a diminished ovarian reserve is the principal factor of poor ovarian response. Several strategies have been proposed for the management of poor responders, including flare up GnRH agonist regimens and the GnRH antagonist, which presents a new hope in this group of patients.

Comparisons: Poor responder patients (see inclusion criteria) commencing an IVF treatment cyle will receive ovarian stimulation treatment either using a GnRH antagonist (Ganirelix) or flare up agonist (Arvekap) protocol. Primary outcomes compared will be ongoing pregnancy rates in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycle
* 1 or more failed IVF attempts with poor response
* 5 or fewer oocytes retrieved
* FSH>12 IU/l on day 3

Exclusion Criteria:

* PCOS
* Normal responders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270
Dates: Start 2003-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate per embryo transfer

SECONDARY OUTCOMES:
Duration of ovarian stimulation, total rFSH used, estradiol, LH and progesterone concentration on hCG day.
Number of mature oocytes retrieved.
Number of fertilised oocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Tarlatzis BC, Zepiridis L, Grimbizis G, Bontis J. Clinical management of low ovarian response to stimulation for IVF: a systematic review. Hum Reprod Update. 2003 Jan-Feb;9(1):61-76. doi: 10.1093/humupd/dmg007. PMID 12638782
- [Derived] Lainas TG, Sfontouris IA, Papanikolaou EG, Zorzovilis JZ, Petsas GK, Lainas GT, Kolibianakis EM. Flexible GnRH antagonist versus flare-up GnRH agonist protocol in poor responders treated by IVF: a randomized controlled trial. Hum Reprod. 2008 Jun;23(6):1355-8. doi: 10.1093/humrep/den107. Epub 2008 Apr 10. PMID 18403419